CLINICAL TRIAL: NCT05407441
Title: TAZNI: A Phase I/II Combination Trial of Tazemetostat With Nivolumab and Ipilimumab for Children With INI1-Negative or SMARCA4-Deficient Tumors
Brief Title: Tazemetostat+Nivo/Ipi in INI1-Neg/SMARCA4-Def Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Susan Chi, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Epizyme, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Susan Chi, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-041
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Atypical Teratoid Rhabdoid Tumor; INI1 (SMARCB1)-Deficient Primary CNS Malignant Tumors; SMARCA4-deficient Primary CNS Malignant Tumors; Malignant Rhabdoid Tumor (MRT); Rhabdoid Tumor of the Kidney (RTK); Epithelioid Sarcoma; Chordoma
Keywords: Atypical Teratoid Rhabdoid Tumor; INI1 (SMARCB1)-deficient primary CNS malignant tumors; SMARCA4-deficient primary CNS malignant tumors; Malignant rhabdoid tumor (MRT); Rhabdoid Tumor of the Kidney (RTK); Epithelioid Sarcoma; Chordoma
MeSH Terms: conditions — Rhabdoid Tumor; Sarcoma; Chordoma | interventions — tazemetostat; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase I a: DOSE ESCALATION (STRATUM A, ATRT and primary CNS malignant tumor, INI/SMARCA4-deficient) (Experimental): Part 1 will be two concurrent "rolling six" phase 1 studies starting at a different tazemetostat dose for each stratum), with one dose escalation and one dose de-escalation planned. All subjects will receive the same nivolumab and ipilimumab doses and dosing schedule
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab
- Phase I b: DOSE ESCALATION (STRATUM B, NON-ATRT, NON-CNS) (Experimental): Part 1 will be two concurrent "rolling six" phase 1 studies starting at a different tazemetostat dose for each stratum), with one dose escalation and one dose de-escalation planned. All subjects will receive the same nivolumab and ipilimumab doses and dosing schedule
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab
- EXP A1: TAZEMETOSTAT + NIVOLUMAB + IPILIMUMAB DOSE EXPANSION (SUBSTRATA A1) (Experimental): Once the MTD or RP2D of the combination is determined for each stratum, the Part 2 portion will open for that stratum, with subjects from Part 1 who are treated at the RP2D to be counted towards the enrollment numbers for Part 2.
  Part 2 will consist of 3 substrata per stratum based on their disease status
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab
- EXP A2: TAZEMETOSTAT + NIVOLUMAB + IPILIMUMAB DOSE EXPANSION (SUBSTRATA A2) (Experimental): Once the MTD or RP2D of the combination is determined for each stratum, the Part 2 portion will open for that stratum, with subjects from Part 1 who are treated at the RP2D to be counted towards the enrollment numbers for Part 2.
  Part 2 will consist of 3 substrata per stratum based on their disease status
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab
- EXP A3: TAZEMETOSTAT + NIVOLUMAB + IPILIMUMAB DOSE EXPANSION (SUBSTRATA A3) (Experimental): Once the MTD or RP2D of the combination is determined for each stratum, the Part 2 portion will open for that stratum, with subjects from Part 1 who are treated at the RP2D to be counted towards the enrollment numbers for Part 2.
  Part 2 will consist of 3 substrata per stratum based on their disease status
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab
- EXP B1: TAZEMETOSTAT + NIVOLUMAB + IPILIMUMAB DOSE EXPANSION (SUBSTRATA B1) (Experimental): Once the MTD or RP2D of the combination is determined for each stratum, the Part 2 portion will open for that stratum, with subjects from Part 1 who are treated at the RP2D to be counted towards the enrollment numbers for Part 2.
  Part 2 will consist of 3 substrata per stratum based on their disease status
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab
- EXP B2: TAZEMETOSTAT + NIVOLUMAB + IPILIMUMAB DOSE EXPANSION (SUBSTRATA B2) (Experimental): Once the MTD or RP2D of the combination is determined for each stratum, the Part 2 portion will open for that stratum, with subjects from Part 1 who are treated at the RP2D to be counted towards the enrollment numbers for Part 2.
  Part 2 will consist of 3 substrata per stratum based on their disease status
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab
- EXP B3: TAZEMETOSTAT + NIVOLUMAB + IPILIMUMAB DOSE EXPANSION (SUBSTRATA B3) (Experimental): Once the MTD or RP2D of the combination is determined for each stratum, the Part 2 portion will open for that stratum, with subjects from Part 1 who are treated at the RP2D to be counted towards the enrollment numbers for Part 2.
  Part 2 will consist of 3 substrata per stratum based on their disease status
  Interventions: Drug: Tazemetostat; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Tazemetostat — oral, twice daily, dosage per protocol
  Other Names: TAZVERIK
Drug: Nivolumab — IV, dosage and schedule per protocol
  Other Names: OPDIVO
Drug: Ipilimumab — IV, dosage and schedule per protocol
  Other Names: YERVOY

SUMMARY:
This research study involves a combination of three drugs given together as a possible treatment for malignant rhabdoid tumor, atypical teratoid rhabdoid tumor, epithelioid sarcoma, chordoma or other tumors that are deficient in one of two possible proteins, either INI-1 (SMARCB1) or SMARCA4.

The names of the study drugs involved in this study are:

* Tazemetostat (TAZVERIK)
* Nivolumab (OPDIVO)
* Ipilimumab (YERVOY)

DETAILED DESCRIPTION:
This research study involves a combination of three drugs given together as a possible treatment for these types of cancers. One drug is small molecule inhibitor targeting EZH2 (tazemetostat) and two are immunotherapeutic checkpoint inhibitors (nivolumab and ipilimumab). This is a Phase I/II clinical trial. Phase I clinical trials test the safety of an investigational drug, or combination of drugs, and tries to define the appropriate dose of the investigational drugs to use for further studies. Phase II clinical trials test the safety and effectiveness of an investigational drug, or drug combination, to learn whether the drug or drug combination works in treating a specific disease. "Investigational" means that the drug combination is being studied.

This trial is studying the combination of tazemetostat, nivolumab, and ipilimumab in two parts:

* Part 1: To find the safest dose of these three study drugs in combination for children with INI1- (or SMARCA4-) negative cancers who have completed upfront treatment
* Part 2: To determine whether this combination can effectively treat INI1- or SMARCA4-negative cancers

The research study procedures include screening for eligibility study treatment, evaluation and follow-up visits. Participants will be asked to provide blood samples and undergo procedures that might be different from a regular medical examination. There are additional research samples that participants will be asked to consent for their collection.

Participants will receive study treatment for up to 2 years, as long as there is benefit or there are no serious side effects. Participants will be followed for approximately 2 years after stopping treatment.

It is expected that about 49 people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has not approved this combination of three drugs for this specific disease. However, tazemetostat has been approved for use in epithelioid sarcoma (an INI1-deficient tumor), and the combination of nivolumab and ipilimumab has also been approved for other uses. Separately, tazemetostat and the combination of nivolumab and ipilimumab have also been tested in children and the safest doses of each drug (and the combination for nivolumab and ipilimumab) have been determined.

Bristol-Myers Squibb and Epizyme, two pharmaceutical companies, are supporting this study by providing the study drugs. Dana-Farber Cancer Institute is also supporting this study by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed tumors at diagnosis or at relapse (as applicable):
* Stratum A

  * Atypical Teratoid Rhabdoid Tumor (ATRT)
  * Other INI1- or SMARCA4-deficient primary CNS malignant tumors (with PI approval)
* Stratum B

  * Malignant rhabdoid tumor (MRT)
  * Rhabdoid tumor of the kidney (RTK)
  * Epithelioid sarcoma
  * Chordoma (poorly differentiated or de-differentiated)
  * Other INI1- or SMARCA4-deficient malignant tumors (with PI approval)
* All subjects must have had tumor assessment at original diagnosis or relapse showing either of the following: Loss of INI1 confirmed by immunohistochemistry (IHC) OR molecular confirmation of tumor bi-allelic SMARCB1 (INI1) loss or mutation when INI1 IHC is equivocal or unavailable
* Loss of SMARCA4 confirmed by IHC OR molecular confirmation of tumor SMARCA4 loss or mutation (with PI approval) Reports confirming these findings (including tumor sequencing if available) will be reviewed by the Sponsor-Investigator, PI or designee for approval of eligibility prior to enrollment.
* Treatment status: All subjects must have completed planned upfront treatment for their disease for strata A1 or B1. Subjects need not have relapsed or have refractory disease to be eligible for this protocol.
* Disease Status: For subjects under consideration for strata A1 or B1, subjects must have evaluable disease Note: Leptomeningeal lesions/disease are allowed as evaluable disease.
* For relapsed/refractory subjects under consideration for strata A2 or B2, subjects must have measurable disease as defined by RANO for stratum A2 or RECIST v1.1 for stratum B2. See Section 11.
* Note: the following do not qualify as measurable disease:

  * malignant fluid collections (e.g., ascites, pleural effusions)
  * bone marrow infiltration
  * lesions only detected by nuclear medicine studies (e.g., bone, gallium or PET scans)
  * elevated tumor markers in plasma or CSF
  * previously irradiated lesions that have not demonstrated clear progression post- radiation therapy
  * leptomeningeal lesions that do not meet the measurement requirements for RANO.
* For subjects under consideration for strata A3 or B3, subjects must have no evidence of evaluable or measurable disease by exam or imaging.
* Pre-recurrent subjects to be enrolled in strata A1, B1, A3, or B3 must be enrolled within 8 weeks of completion of upfront therapy
* Age ≥ 6 months and ≤ 21years of age
* Karnofsky performance status ≥ 50% for subjects ≥16 years of age and Lansky performance status ≥ 50% for subjects <16 years of age (see Appendix A). Note: Neurologic deficits in subjects with CNS tumors must have been stable for at least 7 days prior to study enrollment. Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Life expectancy of greater than 2 months.
* Prior Therapy: Subjects must have fully recovered from the acute toxic effects of all prior anti-cancer therapy. Subjects must meet the following minimum washout periods prior to first day of study treatment:

  * Myelosuppressive chemotherapy: ≥21 days after the last dose of myelosuppressive chemotherapy.
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or ANC counts): ≥ 7 days after the last dose of the agent.
  * Small molecule biologic therapy: ≥7 days following the last dose of a non-monoclonal biologic agent.
  * Monoclonal antibody: ≥21 days after the last dose, and toxicity related to prior antibody therapy must be recovered to Grade ≤1.
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid. CNS subjects receiving corticosteroids for neurologic symptom relief must be at stable or decreasing doses for at least 7 days prior to the first day of study treatment. For all patients, corticosteroid doses of up to 0.12 mg/kg/day prednisone equivalent may be approved after consultation with the Principal Investigator. Treatment with topical, inhaled or ophthalmic corticosteroid is acceptable.
* Radiotherapy

  * ≥14 days after focal XRT (small port)
  * ≥90 days must have elapsed after prior TBI, craniospinal XRT or if >50% irradiation of pelvis
  * ≥42 days must have elapsed if other substantial bone marrow irradiation
  * ≥42 days must have passed since last radionuclide therapy (e.g. samarium or radium).
  * Myeloid growth factors: ≥14 days following the last dose of long-acting growth factor (e.g. Neulasta) or 7 days following short-acting growth factor.
  * Autologous stem cell therapy, Autologous T Cell, or other CellularTherapy: ≥ 42 days must have elapsed after any cellular therapy infusion. Prior allogeneic stem cell transplant is not allowable.
  * Prior EZH2 inhibitor therapy: Subjects with relapsed/refractory disease (strata A2 and B2) may have received prior single agent tazemetostat or other EZH2 inhibitors for up to 1 year, but subjects without prior progression/relapse may NOT have received any prior EZH2 inhibitors.
* Subjects must have adequate organ function as defined below:

  * Bone Marrow Function
  * Absolute neutrophil count ≥1,000/uL
  * Hemoglobin ≥8 g/dL (may receive RBC transfusions)
  * Platelets: For non-relapsed subjects (Strata A1, A3, B1 or B3): >75K/uL, For subjects with relapsed disease (Strata A2 or B2): >50K/uL, For all subjects: must be platelet transfusion independent, defined as not receiving a platelet transfusion for at least 7 days prior to CBC documenting eligibility.
* Hepatic Function

  * Total bilirubin ≤ 1.5 x upper limit of normal for age.
  * ALT (SGPT) and AST (SGOT) ≤ 3 x upper limit of normal (for the purpose of this study, the ULN for ALT is 45 U/L)
* Renal Function: A serum creatinine based on age/gender as follows: Maximum Serum Creatinine (mg/dL)

  * Male: 6 months to 1 year-0.5,1 to < 2 years-0.6, 2 to < 6 years-0.8, 6 to < 10 years-1, 10 to < 13 years-1.2,13 to < 16 years- 1.5, ≥ 16 years 1.7
  * Female: 6 months to 1 year-0.5,1 to < 2 years-0.6, 2 to < 6 years-0.8, 6 to < 10 years-1, 10 to < 13 years-1.2,13 to < 16 years- 1.4, ≥ 16 years1.4 OR
  * Creatinine clearance ≥ 70 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Adequate Pulmonary Function defined as: No evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficient and a pulse oximetry > 92% while breathing room air.

  -- Adequate Neurologic Function defined as: Subjects with seizure disorder may be enrolled if on anticonvulsants and well controlled. Nervous system disorders (CTCAE v5.0) resulting from prior therapy must be ≤ Grade 2, with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible.
* Negative B-HCG pregnancy test (urine or serum) in females of childbearing potential.
* Women of childbearing potential (WOCBP) receiving the TAZNI combination agree to adhere to contraception for a period of 5 months after the last dose of either tazemetostat, nivolumab, or ipilimumab
* Men receiving the TAZNI combination and who are sexually active with WOCBP will agree to adhere to barrier contraception for a period of 3 months after the last dose of either tazemetostat, nivolumab or ipilimumab.
* Ability to understand and/or the willingness of the subject (or parent or legally authorized representative, if minor) to provide informed consent, documented using an institutionally approved informed consent procedure.

Exclusion Criteria:

* Concomitant Medications
* Subjects who are receiving any other investigational agents or other anti-cancer agents are not eligible.
* CYP3A4 Agents: Subjects who are currently receiving drugs that are strong or moderate inducers or inhibitors of CYP3A4 are not eligible. Such inducers or inhibitors of CYP3A4 are prohibited from 14 days prior to the first dose of tazemetostat to the end of the study. See Appendix C for a list of agents. Note:Dexamethasone for CNS tumors or metastases, on a stable or decreasing dose, is allowed up to 0.12mg/kg/day prednisone equivalents.
* Subjects with a known history of HIV, hepatitis B, and/or hepatitis C (testing not required as part of screening).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or any other concurrent disease which in the judgment of the Investigator would make the subject inappropriate for enrollment on this study.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has active autoimmune disease that has required systemic treatment in the past 12 months, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are exceptions. Intermittent use of bronchodilators or local steroid injections are not excluded. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Autoimmune diagnoses not listed must be approved by the Principal Investigator.
* On screening CBC differential, subjects must not have any significant morphologic abnormalities concerning for MPN/MDS or ALL.
* Subjects must not have any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS) or prior history of lymphoblastic lymphoma (LBL) or leukemia (ALL).
* Subjects who have received prior solid organ transplantation are not eligible.
* Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as there is yet no available information regarding human fetal or teratogenic toxicities.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA4 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. OX40, CD137).
* Subjects who have received live / attenuated vaccine within 30 days of first dose of study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tazemetostat or Orasweet.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3 or Higher Treatment-Related Toxicity | AE to be collected continuously after the patient has provided informed consent through up to 30 days after last dose of study treatment up to 5.5 years
  All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAE v5 as reported on case report forms will be counted. Incidence is the number of patients experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.
Maximal Tolerated Dose (MTD) | Treatment duration is a median of N cycles range (t1 - t2). Treatment continues until disease progression or unacceptable toxicity up to 5.5 years
  The MTD defined as the dose level associated with observed DLTs in <33% of enrolled subjects. The DLT assessment will be restricted to the first cycle.

SECONDARY OUTCOMES:
Recommended Pediatric Phase 2 Dose (RP2D) | Treatment duration is a median of N cycles range (t1 - t2). Treatment continues until disease progression or unacceptable toxicity up to 5.5 years
Overall Response Rate (ORR) | Disease is evaluated each cycle on treatment; Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of N cycles range (t1 - t2) up to 5.5 years
  The objective response rate (ORR) is defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 or RANO criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Median Overall Survival (OS) | Up through 5.5 years
  OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Median Progression-free survival (PFS) | Participants are followed for survival every 6 months, up to 3 years after treatment discontinuation
  Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Roden AC. Molecularly Defined Thoracic Neoplasms. Adv Anat Pathol. 2024 Sep 1;31(5):303-317. doi: 10.1097/PAP.0000000000000439. Epub 2024 Mar 19. PMID 38501690